CLINICAL TRIAL: NCT06049420
Title: Lifestyle Medicine: Establishing Clinical Approaches to Chronic Disease for Rural Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia School of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Christopher Pankey, Associate Professor, West Virginia School of Osteopathic Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R010422CP
Record Dates: First submitted 2023-09-12; First posted 2023-09-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Hyperlipidemias; Polycystic Ovary Syndrome; Hypertension; Coronary Heart Disease; Heart Failure; Depression, Anxiety; Type II Diabetes; Metabolic Syndrome
Keywords: lifestyle; chronic disease; physical activity
MeSH Terms: conditions — Obesity; Hyperlipidemias; Polycystic Ovary Syndrome; Hypertension; Coronary Disease; Heart Failure; Depression; Anxiety Disorders; Diabetes Mellitus, Type 2; Metabolic Syndrome; Chronic Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be able to opt-in to the protocol for adjunctive treatment, and their outcome measures will be assessed relative to similar patients that do not opt-in to the intervention (standard care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): participants that have received a referral, and opt-in for the adjunctive treatment plan
  Interventions: Behavioral: Lifestyle counseling and coaching

INTERVENTIONS:
Behavioral: Lifestyle counseling and coaching — Each participant will be provided with personalized exercise therapy that is best suited for their personal goals and disease states. Participants in this study will be encouraged to establish accountability through setting SMART goals, and through monitoring their activity using wearable fitness technology provided to them. This program will also aim to create a sense of community as group activity classes will be available for those that wish to attend. Individualized exercise/physical activity prescriptions will be provided and discussed.

SUMMARY:
Developed nations worldwide are currently enduring a health crisis, as chronic diseases continue to decrease quality of life and promote additional disease states or even death for much of the population. Rural populations are at a particular disadvantage, as they lack access to health clubs, wellness programs and similar resources that are more available in urban areas. Although pharmaceutical therapies have continued to show therapeutic advancements, the rates of disease onset and death from chronic disease has not seen similar improvements, and in fact continue to worsen. Excitingly, significant evidence has been published demonstrating an affordable, effective treatment to directly treat and prevent these chronic diseases, but few have demonstrated successful implementation of this therapy, which is improved lifestyle. Specifically, physical activity and healthy body composition are powerful therapeutics that have been demonstrated to effectively combat and prevent chronic diseases. Additionally, improving these lifestyle factors are often more effective than pharmaceutical interventions without the wide range of side effects. Unfortunately, barriers exist on multiple tiers in the practice of family medicine that demote the implementation of lifestyle medicine. To better serve patients at risk of, or suffering from chronic disease, the investigators are seeking to establish a lifestyle medicine prescription program for rural West Virginia. This program will provide patient education on the benefits of physical activity, body composition, and help patients identify strategies to implement healthy lifestyle choices that can be sustainable for the long-term. Patients will be advised on local opportunities to increase physical activity (yoga studio, martial arts, fitness facilities, aquatic center, etc.) and provided access to the facilities they are most likely to adhere to regularly. They will also be provided training on exercise techniques, equipment, and facilities to increase familiarity and comfort in these settings.

DETAILED DESCRIPTION:
Patients will have the option to opt-in to this program if they receive a referral from their primary care physician at the Robert C. Byrd Clinic (RCBC). The referral period will be one month long, followed by 3 months of wellness facility access (intervention period). This pilot program will be restricted to adults (18-64 years old) with two or more diagnosed chronic diseases. Program admittance will be restricted to patients with diseases that have sufficient evidence for the efficacy of exercise therapy. As patients will be referred to the program, they will all have physician consent to participate in supervised physical activity. Standard care will proceed as determined by the primary care physician, as this program will be adjunctive treatment. As patient recruitment is contingent on physician referrals, the investigators have established a strong network with the family care physicians and administration from RCBC, and they are very confident that this program will be in high demand. Physicians will be reminded of the recruitment time 1-2 times/month for the 3 months preceding the start date by email, personal communication, and lunch seminars. Prior to accessing the wellness facility, each patient will be scheduled for an intake meeting. This intake meeting will be used to collect patient information (such as vital signs, morphometrics, demographics, physical activity history and readiness, health history, etc.), and understand patient goals (weight loss, glucose management, pain relief, blood pressure management, etc.). A patient questionnaire will be developed for this meeting, and patients will also fill out a physical activity readiness questionnaire. Motivational interviewing techniques will be implemented to promote adherence to the program. Individualized goals will be determined and recorded. Patient preferences such as individual training/coaching vs. group fitness will also be determined. Following the intake meeting, each patient will be advised on how they may best reach their goals, and support will be provided by the PI or a trained medical student for implementation of physical activity. The wellness facility (Greenbrier Valley Fitness) was specifically chosen as it offers a wide variety of exercise equipment and activities including strength training, cross training, group fitness, yoga, and many others. The PI or student research technicians will be present for questions, coaching, and monitoring at all times when the patient is being active. Each patient will be provided with personalized exercise therapy that is best suited for their personal goals and disease states.

An overarching goal is for each patient to achieve 150 minutes per week of moderate to vigorous physical activity. This benchmark was chosen as it is the current recommendation from the CDC [1], and has been demonstrated to be therapeutic for all, and curative for some, of the chronic diseases mentioned above [2,3]. Importantly, some patients may not make this goal within the allotted time-frame depending on their current fitness and disease states. In order to assess adherence and attrition, the investigators will have to assess individuals based on their individualized goals. Any participant that fails to attend >50% of their scheduled activities, or fails to show up at least once in the last 15 days of the study will count as drop-outs.

Data collected on patients will only occur after their referral to our program, so that no patient data will be shared between institutions (WVSOM and the Robert C. Byrd Clinic) and so that the investigators can properly deliver informed consent to patients that are willing to have their data used for research purposes. GraphPad Prism and excel software will be used to store and analyze the data, using the descriptive statistics and computational functions to provide count data and attrition rates. Additional analyses of factors such as disease prevalence, demographics, age, gender, and appropriate interactions may also be assessed contingent on the study population.

ELIGIBILITY:
Inclusion Criteria:

* Program admittance will be restricted to patients with 2+ diagnosed diseases that have sufficient evidence for the efficacy of exercise therapy (obesity, hyperlipidemia, metabolic syndrome, polycystic ovarian syndrome, type II diabetes, hypertension, coronary heart disease, heart failure, depression, anxiety)
* physician referral required

Exclusion Criteria:

* no chronic disease diagnosis, lack of physician referral, unwillingness to participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Demand | 1 month
  initial demand for the program
Attrition rate | 4 months
  Drop out rate after opting in to the intervention
physical activity | 4 months
  minutes of moderate to vigorous physical activity
Body Composition | Once at enrollment, and once at cessation of the intervention 4 weeks later.
  Fat mass (kg) and Fat free mass (kg) will be collected pre- and post-intervention
Body Composition | Once at enrollment, and once at cessation of the intervention 4 weeks later.
  bone mineral content (g) will be collected pre- and post-intervention
Body Composition | Once at enrollment, and once at cessation of the intervention 4 weeks later.
  bone density (g/cm^2)) will be collected pre- and post-intervention

SECONDARY OUTCOMES:
Blood pressure | 4 Months
  Systolic and diastolic blood pressure (mmHg)
Blood glucose | 4 Months
  mg/dL
blood lipids | 4 Months
  triglycerides (mg/dL)
Glycosylated hemoglobin | 4 Months
  A1C (percent of hemoglobin that is glycosylated)
BMI | 4 Months
  weight and height will be combined to report BMI in kg/m^2
total cholesterol | 4 Months
  Triglycerides, High density lipoproteins (HDL) and low density lipoproteins (LDL) will be used to determine total cholesterol.
Self-efficacy | 4 Months
  Exercise Self Efficacy scale - ranges from 0 (low self efficacy) to 10 (high self efficacy)
  These data measure individual's confidence in his or her capacity to execute behaviors necessary to maintain an active lifestyle.
Basal Metabolic Rate | Recordings will occur once at enrollment, and once at the end of the intervention 4 weeks later.
  Metabolic rate will be estimated via indirect calorimetry using a respiratory gas analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Pankey, Ph.D., Principal Investigator — West Virginia School of Osteopathic Medicine
Locations (1):
- West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palakodeti S, Uratsu CS, Schmittdiel JA, Grant RW. Changes in physical activity among adults with diabetes: a longitudinal cohort study of inactive patients with Type 2 diabetes who become physically active. Diabet Med. 2015 Aug;32(8):1051-7. doi: 10.1111/dme.12748. Epub 2015 Apr 10. PMID 25764298
- [Background] Hupin D, Roche F, Gremeaux V, Chatard JC, Oriol M, Gaspoz JM, Barthelemy JC, Edouard P. Even a low-dose of moderate-to-vigorous physical activity reduces mortality by 22% in adults aged >/=60 years: a systematic review and meta-analysis. Br J Sports Med. 2015 Oct;49(19):1262-7. doi: 10.1136/bjsports-2014-094306. Epub 2015 Aug 3. PMID 26238869
- See also: [1] CDC. Physical Activity. Centers for Disease Control and Prevention. Published July 25, 2022. Accessed October 7, 2022. — https://www.cdc.gov/physicalactivity/index.html